CLINICAL TRIAL: NCT00511160
Title: Prevalence of Cardiotropic Viruses in Cardiac Surgery Patients Without Clinical Evidence of Myocarditis or Myocarditic Sequelae
Brief Title: Cardiotropic Viruses in Cardiac Surgery Patients Without Clinical Evidence of Myocarditis or Myocarditic Sequelae
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to logistical/personnel difficulties
Sponsor: Udo Sechtem (Other)
Responsible Party: Sponsor-Investigator, Udo Sechtem, Prof. Udo Sechtem, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Organization: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: RBK103
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Myocarditis
Keywords: myocarditis; parvovirus B19 (PVB19); human herpes virus 6 (HHV6); cardiac magnetic resonance tomography (CMR)
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S (Active Comparator): Study arm: Cardiac surgery group
  Interventions: Procedure: Myocardial biopsies with TRU CUT 14 Gauge needle
- C (Active Comparator): Routine cardiology group
  Interventions: Procedure: Endomyocardial biopsies

INTERVENTIONS:
Procedure: Myocardial biopsies with TRU CUT 14 Gauge needle — Myocardial needle biopsy and right atrial appendectomy
  Other Names: TRU CUT 14 Gauge needle
  Arms: S
Procedure: Endomyocardial biopsies — The control arm C consists of routine-workup of patients with suspected myocarditis, independent of the study arm C, but with analogous screening methods and comparable biopsy sampling
  Arms: C

SUMMARY:
Myocarditis is mainly caused by cardiotropic viruses. In recent time viruses found in endomyocardial biopsies mainly consist of parvovirus B19 (PVB19) and human herpesvirus 6 (HHV6). A definite causal link between virus-genome detection of PVB19 and/or HHV6 (via pcr techniques)and cardiac inflammation and dysfunction is however still missing.

Primary objective:

To determine the prevalence of PVB19 and HHV6 virus genome in heart muscle biopsies of cardiac surgery patients without clinical evidence of myocarditis or myocarditic sequelae

Secondary objectives:

1. Correlation of non-invasive myocarditis screening exams (cardiac magnetic resonance, ecg, history, inflammatory markers) with biopsy results
2. Prognostic value of virus prevalence for the postoperative course

Primary hypothesis:

Patients without clinical evidence of myocarditis or myocarditic sequelae demonstrate to a significant lesser extent inflammatory activity and virus genome in their myocardium as compared to patients being clinical suspicious for myocarditis.

DETAILED DESCRIPTION:
Prospective monocentric study with to 2 arms

Study arm: Cardiac surgery group, Control arm: Routine cardiology group Minimum of 100 patients included into the study arm

Inclusion criteria for the study arm:

Adult patients having cardiac surgery done under use of cardiopulmonary bypass

Data collection:

Past medical history, ecg, prior cardiovascular imaging (echo, ventriculography), cardiac magnetic resonance imaging (CMR), serologic studies, work-up of endomyocardial biopsies (histology, molecular-pathology, follow-up CMR.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* No ability to give informed consent
* presence of so far accepted parvovirus/herpesvirus associated comorbidities
* contraindications for magnetic resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine the prevalence of PVB19 and HHV6 virus genome in heart muscle biopsies of cardiac surgery patients without clinical evidence of myocarditis or myocarditic sequelae | 2 years

SECONDARY OUTCOMES:
Correlation of non-invasive myocarditis screening exams (cardiac magnetic resonance, ecg, history, inflammatory markers) with biopsy results | 2 years
Prognostic value of virus prevalence for the postoperative course | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Udo P Sechtem, MD, Study Chair — Head of Cardiology, Robert Bosch Krankenhaus, Stuttgart, Germany; Ulrich FW Franke, MD, Study Director — Head of Cardiovascular Surgery, Robert Bosch Krankenhaus, Stuttgart, Germany; Reinhardt Kandolf, MD, Study Director — Director of Institute of Molecular Pathology University Tuebingen, Germany; Hannibal Baccouche, MD, Principal Investigator — Department of Cardiology, Robert Bosch Krankenhaus, Stuttgart, Germany; Hardy Baumbach, MD, Principal Investigator — Department of Cardiovascular Surgery, Robert Bosch Krankenhaus Stuttgart, Germany
Locations (1):
- Robert Bosch Krankenhaus, Auerbachstrasse 110, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No